CLINICAL TRIAL: NCT02153177
Title: The Effect of NSAIDs After a Rotator Cuff Repair Surgery. A Prospective Randomized Controlled Trial
Brief Title: The Effect of NSAIDs After a Rotator Cuff Repair Surgery.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was withdrawn prior to any participants being enrolled.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB 14-0540
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Rotator Cuff Tear
Keywords: Randomized Controlled Trial (RCT); RCT; rotator cuff tear; NSAIDs; non-steroidal anti-inflammatory drugs; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Ibuprofen; Hydrocodone; Acetaminophen; Omeprazole; oxycodone-acetaminophen

ARMS (2):
- NSAID and pain medication arm (Active Comparator): After a rotator cuff repair procedure subjects in the NSAID and pain medication arm will receive both Ibuprofen and Hydrocodone/Acetaminophen, and also Omeprazole.
  Interventions: Procedure: Rotator cuff repair; Drug: Ibuprofen, Hydrocodone/Acetaminophen, Omeprazole
- pain medication arm (Active Comparator): Patients in the pain medication arm will receive Hydrocodone/Acetaminophen after the rotator cuff repair procedure.
  Interventions: Procedure: Rotator cuff repair; Drug: Hydrocodone/Acetaminophen

INTERVENTIONS:
Procedure: Rotator cuff repair — Arthroscopic procedure
  Other Names: Rotator cuff repair procedure
Drug: Ibuprofen, Hydrocodone/Acetaminophen, Omeprazole — In addition to pain medication after the procedure patients will receive Ibuprofen and Omeprazole. Omeprazole is given to minimize the gastrointestinal side effects of Ibuprofen.
  Other Names: Motrin, Advil (Ibuprofen); Norco (Hydrocodone/Acetaminophen); Prilosec (Omeprazole)
  Arms: NSAID and pain medication arm
Drug: Hydrocodone/Acetaminophen — Hydrocodone/Acetaminophen is given for pain control after the surgery.
  Other Names: Norco
  Arms: pain medication arm

SUMMARY:
The main purpose of the study is to determine the effect of Non-steroidal Anti-inflammatory Drugs (NSAIDs) on the healing process after a rotator cuff repair procedure.

DETAILED DESCRIPTION:
Furthermore, the study will also determine the rate of narcotic medications use and the retear rate after a rotator cuff repair procedure.

ELIGIBILITY:
Inclusion Criteria:

* rotator cuff tear
* age 45-75 years

Exclusion Criteria:

* diabetes
* pregnancy
* chronic kidney disease
* liver cirrhosis
* hematologic malignancy
* alcohol abusing
* drug abusing

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | one year
  The scale measures pain from 0 to 10 and also includes a questionnaire for assessing the activity of daily living.

SECONDARY OUTCOMES:
Ultrasound evaluation of retear rate | one year
  Ultrasound evaluation of retear rate at 6 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lewis L Shi, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States